CLINICAL TRIAL: NCT00244244
Title: A Multicenter, Dose Ranging Safety and Pharmacokinetics Study of Arimoclomol in Amyotrophic Lateral Sclerosis (ALS)
Brief Title: A Multicenter, Dose Ranging Safety and Pharmacokinetics Study of Arimoclomol in ALS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CytRx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: AALS-001
Record Dates: First submitted 2005-10-25; First posted 2005-10-26 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — arimoclomol

INTERVENTIONS:
Drug: arimoclomol

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability of arimoclomol in ALS patients following 90 days of dosing. In addition, the amount of arimoclomol in blood and cerebrospinal fluid will be measured.

DETAILED DESCRIPTION:
Arimoclomol is a small molecule that upregulates "molecular chaperones" in cells under stress. Arimoclomol extends survival by five weeks when given both pre-symptomatically and at disease onset in a mutant superoxide dismutase (SOD1) transgenic mouse model of ALS. Furthermore, it has been demonstrated to have neuroprotective and neuroregenerative effects in other rat models of nerve damage. Molecular chaperone proteins are critical in the cellular response to stress and protein misfolding. Recent data suggest that the SOD1 mutation responsible for ALS in some patients with familial disease reduces the availability of a variety of molecular chaperones, and thus weakens their ability to respond to cellular stress. Protein misfolding and consequent aggregation may play a role in the pathogenesis of both the familial and sporadic forms of ALS. Therapeutic agents such as arimoclomol that improve cellular chaperone response to protein misfolding may be helpful in ALS.

ELIGIBILITY:
Inclusion Criteria:

* Familial or sporadic ALS
* Vital capacity equal to or more than 60% predicted value for gender, height and age at the screening visit
* First ALS symptoms occurred no more than five years prior to screening
* Must be able to take oral medication

Exclusion Criteria:

* Dependence on mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2005-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Safety

SECONDARY OUTCOMES:
Pharmacokinetics
ALSFRS-R
Vital Capacity

CONTACTS AND LOCATIONS:
Overall Officials: Merit Cudkowicz, MD, Principal Investigator — Massachusetts General Hospital; Jeremy Shefner, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (10):
- United States (10):
  - University of California, Irvine Medical Center, Irvine, California
  - University of Miami School of Medicine, Miami, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Hennepin Faculty Associates/Berman Center, Minneapolis, Minnesota
  - SUNY Upstate Medical University, Syracuse, New York
  - Duke University, Durham, North Carolina
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Background] Kieran D, Kalmar B, Dick JR, Riddoch-Contreras J, Burnstock G, Greensmith L. Treatment with arimoclomol, a coinducer of heat shock proteins, delays disease progression in ALS mice. Nat Med. 2004 Apr;10(4):402-5. doi: 10.1038/nm1021. Epub 2004 Mar 21. PMID 15034571
- [Background] Benn SC, Brown RH Jr. Putting the heat on ALS. Nat Med. 2004 Apr;10(4):345-7. doi: 10.1038/nm0404-345. No abstract available. PMID 15057226
- [Background] Kurthy M, Mogyorosi T, Nagy K, Kukorelli T, Jednakovits A, Talosi L, Biro K. Effect of BRX-220 against peripheral neuropathy and insulin resistance in diabetic rat models. Ann N Y Acad Sci. 2002 Jun;967:482-9. doi: 10.1111/j.1749-6632.2002.tb04306.x. PMID 12079878
- [Background] Kalmar B, Burnstock G, Vrbova G, Urbanics R, Csermely P, Greensmith L. Upregulation of heat shock proteins rescues motoneurones from axotomy-induced cell death in neonatal rats. Exp Neurol. 2002 Jul;176(1):87-97. doi: 10.1006/exnr.2002.7945. PMID 12093085
- [Background] Muchowski PJ, Wacker JL. Modulation of neurodegeneration by molecular chaperones. Nat Rev Neurosci. 2005 Jan;6(1):11-22. doi: 10.1038/nrn1587. PMID 15611723
- [Background] Kalmar B, Greensmith L, Malcangio M, McMahon SB, Csermely P, Burnstock G. The effect of treatment with BRX-220, a co-inducer of heat shock proteins, on sensory fibers of the rat following peripheral nerve injury. Exp Neurol. 2003 Dec;184(2):636-47. doi: 10.1016/S0014-4886(03)00343-1. PMID 14769355